CLINICAL TRIAL: NCT02760615
Title: An Open-Label, 2-Part, Multicenter, Post-marketing Study to Evaluate the Effect of Moderately or Severely Active Ulcerative Colitis or Crohn's Disease on Cytochrome P-450 Enzyme Substrates Compared to Healthy Subjects and the Effect of Vedolizumab Treatment on Cytochrome P-450 Enzyme Substrates in Subjects With Ulcerative Colitis or Crohn's Disease
Brief Title: Phase 4, Vedolizumab-4002 Post-marketing, Disease-Drug-Drug Interaction Study
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No enrollment
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Vedolizumab-4002; U1111-1171-3187 (Registry Identifier: WHO)
Record Dates: First submitted 2016-05-02; First posted 2016-05-03 (Estimated); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Colitis, Ulcerative; Crohn Disease
Keywords: Drug therapy
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease | interventions — Caffeine; Losartan; Omeprazole; Dextromethorphan; Midazolam; vedolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: UC and CD Participants (Other): Participants with UC or CD and not concurrently treated with vedolizumab or other biologics will receive caffeine 200 milligram (mg), tablets, orally, once, losartan 50 mg, tablets, orally, once, omeprazole 40 mg, capsules, orally, once, dextromethorphan, 30 mg (2*15 mg), capsules, orally, once, and midazolam 10 mg, syrup, orally, once, on Day 1.
  Interventions: Drug: Caffeine; Drug: Losartan; Drug: Omeprazole; Drug: Dextromethorphan; Drug: Midazolam; Drug: Vedolizumab
- Part 1: Healthy Participants (Other): Healthy participants will receive caffeine 200 mg, tablets, orally, once, losartan 50 mg, tablets, orally, once, omeprazole 40 mg, capsules, orally, once, dextromethorphan 30 mg (2*15 mg), capsules, orally, once, and midazolam 10 mg, syrup, orally, once, on Day 1.
  Interventions: Drug: Caffeine; Drug: Losartan; Drug: Omeprazole; Drug: Dextromethorphan; Drug: Midazolam; Drug: Vedolizumab
- Part 2: Vedolizumab (Experimental): Participants who are on established vedolizumab intravenous (IV) maintenance treatment of 300 mg for treatment of UC or CD and in clinical remission will receive vedolizumab 300 mg IV infusion, once, caffeine 200 mg, tablets, orally, once, losartan 50 mg, tablets, orally, once, omeprazole 40 mg, capsules, orally, once, dextromethorphan 30 mg (2*15 mg), capsules, orally, once, and midazolam 10 mg, syrup, orally, once, on Day 1.
  Interventions: Drug: Caffeine; Drug: Losartan; Drug: Omeprazole; Drug: Dextromethorphan; Drug: Midazolam; Drug: Vedolizumab

INTERVENTIONS:
Drug: Caffeine — Caffeine tablets
Drug: Losartan — Losartan tablets
  Other Names: Cozaar
Drug: Omeprazole — Omeprazole capsules
  Other Names: Prilosec
Drug: Dextromethorphan — Dextromethorphan capsules
  Other Names: Delsym
Drug: Midazolam — Midazolam syrup
  Other Names: Versed
Drug: Vedolizumab — Vedolizumab solution for IV infusion

SUMMARY:
The purpose of this study is to evaluate in a step-wise approach the disease drug-drug interaction (DDI) potential for vedolizumab to indirectly affect the exposure of cytochrome P-450 (CYP) substrate drugs by modulating pro-inflammatory cytokines in participants with ulcerative colitis (UC) or Crohn's disease (CD) who are treated with vedolizumab.

DETAILED DESCRIPTION:
The drug being tested in this study is called vedolizumab, which is being tested to assess the possibility of drug-drug interactions when administered with other medications. The study will comprise of 2 parallel parts: Part 1 and Part 2.

Part 1 will enroll approximately 40 participants: 20 healthy participants and 20 participants with UC or CD who are not currently being treated with vedolizumab. All participants will receive the following medications:

* Caffeine 100 mg
* Losartan 50 mg
* Omeprazole 20 mg
* Dextromethorphan 30 mg
* Midazolam 2 mg

Part 2 will enroll approximately 20 participants on established vedolizumab intravenous (IV) maintenance treatment of 300 mg for the treatment of UC or CD. Participants will receive the same medications and dosages as in Part 1 in addition to their scheduled vedolizumab 300 mg IV.

This multi-center trial will be conducted in the United States. For Part 1 and Part 2, participants will arrive at study unit for check-in (Day -1) and will return to the study unit for dosing and PK assessment on Day 1 and study exit on Day 2 or will be kept from Check-in through at least 24 hours after dosing for safety and PK assessments before discharge. The total confinement period (optional) will be up to 3 days for both the parts. The overall time to participate for each participant in Part 1 will be approximately 6 weeks and for Part 2, it will be approximately 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures including requesting that a participant fast for any laboratory evaluations.
3. Is a cytochrome P-450 (CYP)2C9, CYP2C19, and CYP2D6 extensive metabolizer, based on genotyping of pharmacogenomic (PGx) deoxyribonucleic acid (DNA) analysis.
4. Is a male or female aged 18 to 55 years, inclusive, at Screening.
5. Weighs at least 50 kilogram (kg) and has a body mass index (BMI) of 18.0 to 30 kilogram per square meter (kg/m^2), inclusive, at Screening and Check-in (Day -1).
6. The healthy control participants in Part 1 of this study will be matched at Day-1 with the UC or CD participants in Group 1 or 3 (whichever enrolls faster) on the basis of age (+/-10 years), gender and weight (+/-30 [percent] %).
7. Participants in Part 2 and Group 1 will be matched on Day-1 on the basis of the inflammatory bowel disease (IBD) diagnosis (UC or CD), age (+/-10 years), gender and weight (+/-30%).

   For Part 1 Participants:
8. A male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study.
9. All female participants who are of childbearing potential and who are sexually active, agree to routinely use adequate contraception from signing of informed consent throughout the duration of the study. NOTE: Female participants NOT of childbearing potential are defined as those who have been surgically sterilized (hysterectomy, bilateral oophorectomy, tubal ligation [at least 2 years post-operation]) or who are postmenopausal (example, defined as at least 1 year since last regular menses with an follicle stimulated hormone [FSH] greater than [>] 40 international units per liter [IU/L] or at least 5 years since last regular menses, confirmed before any study medication is implemented).

   For Part 1 Only Participants with UC or CD
10. Has a diagnosis of UC or CD established at least 6 months prior to enrollment by clinical and endoscopic evidence and corroborated by a histopathology report.
11. Prior to entering the study, participants with UC must have had an endoscopy during screening to confirm active disease, with Mayo score of 6 to 12 and an endoscopic subscore greater than or equal to (>=)2. Participants with CD must have a Crohn's Disease Activity Index (CDAI) score of 220 to 450 to confirm moderate to severe disease on entry (that is, Day-1).
12. Participant may be receiving a therapeutic dose of the following drugs for treatment of their underlying disease:

    * Oral or topical 5-aminosalicylic acid (5-ASA) compounds provided that the dose has been stable for the 2 weeks immediately prior to enrollment.
    * Probiotics (example, Culturelle, Saccharomyces boulardii) provided that the dose has been stable for the 2 weeks immediately prior to enrollment.
    * Antidiarrheals (example, loperamide, diphenoxylate with atropine) for control of chronic diarrhea.
    * Azathioprine or 6-mercaptopurine, provided that the dose has been stable for the 8 weeks immediately prior to enrollment.
    * Methotrexate provided that the dose has been stable for the 8 weeks immediately prior to randomization.
    * Oral corticosteroid therapy (prednisone at a stable dose less than or equal to [<=] 30 milligram per day [mg/day], or equivalent steroid) provided that the dose has been stable for the 4 weeks immediately prior to enrollment, if corticosteroids have been initiated, or for the 2 weeks immediately prior to the enrollment, if corticosteroids are being tapered.
13. C-reactive protein (CRP) >=5 milligram per liter (mg/L) during screening period in participants with CD.

    For Part 1 Healthy Participants Only:
14. The participant, in opinion of the investigator, is in healthy condition as determined by a prestudy physical examination, medical history, vital signs, electrocardiogram (ECG), and the results of blood biochemistry, hematology, serology, and urinalysis tests.

    For Part 2 Participants with Active UC and CD:
15. A male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 57 days after last dose.
16. All female participants who are of childbearing potential and who are sexually active with a nonsterilized male partner, agree to routinely use adequate contraception from Screening until 57 days after receiving the last dose of study medication. NOTE: Female participants NOT of childbearing potential are defined as those who have been surgically sterilized (hysterectomy, bilateral oophorectomy, tubal ligation [at least 2 years post-operation]) or who are postmenopausal (example, defined as at least 1 year since last regular menses with an FSH >40 IU/L or at least 5 years since last regular menses, confirmed before any study medication is implemented.
17. Has a diagnosis of UC or CD established at least 6 months prior to enrollment by clinical and endoscopic evidence and corroborated by a histopathology report.
18. Is on established vedolizumab intravenous (IV) for treatment of UC or CD and is in clinical remission as assessed within 7 days of dosing defined for UC; A complete Mayo score of <=2 points and no individual subscore >1 point. For CD; CDAI of <=150 points.
19. Participant may be receiving a therapeutic dose of the following drugs for treatment of their underlying disease:

    * Oral or topical ASA compounds provided that the dose has been stable for the 2 weeks immediately prior to enrollment.
    * Probiotics (example, Culturelle, S. boulardii) provided that the dose has been stable for the 2 weeks immediately prior to enrollment.
    * Antidiarrheals (eg, loperamide, diphenoxylate with atropine) for control of chronic diarrhea.
    * Azathioprine or 6-mercaptopurine, provided that the dose has been stable for the 8 weeks immediately prior to enrollment.
    * Methotrexate provided that the dose has been stable for the 8 weeks immediately prior to randomization.
    * Oral corticosteroid therapy (prednisone at a stable dose <30 mg/day, or equivalent steroid) provided that the dose has been stable for the 4 weeks immediately prior to enrollment if corticosteroids have been initiated or for the 2 weeks immediately prior to the enrollment if corticosteroids are being tapered.

Exclusion Criteria:

For both Part 1 and Part 2:

1. Has a known hypersensitivity to any of the drugs or components in the Injection (Inje) Cocktail.
2. Is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in the conduct of this study (example, spouse, parent, child, sibling) or may consent under duress.
3. Within 30 days prior to enrollment, participants with UC or CD have received any treatment of underlying disease other than those specifically listed in the protocol for the Treatment of UC or CD.
4. If female, the participant is pregnant or lactating or intending to become pregnant before, during, or within 57 days after participating in this study; or intending to donate ova during such time period.
5. If male, the participant intends to donate sperm during the course of this study or for 57 days thereafter.
6. Has received rituximab or natalizumab treatment or other integrin inhibitors.
7. Has taken any excluded medication, supplements, or food products listed in the protocol.
8. Has evidence of abdominal abscess or toxic megacolon at the initial Screening Visit.
9. Has had extensive colonic resection, subtotal or total colectomy.
10. Has had ileostomy, colostomy, or known fixed symptomatic stenosis of the intestine.
11. Has evidence of or has had treatment for Clostridium difficile infection within 60 days or other intestinal pathogen within 30 days prior to enrollment.
12. Has a history or evidence of adenomatous colonic polyps that have not been removed.
13. Has a history or evidence of colonic mucosal dysplasia.
14. Has chronic hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
15. Has any identified congenital or acquired immunodeficiency (example, common variable immunodeficiency, human immunodeficiency virus [HIV] infection, organ transplantation).
16. Has received any live vaccinations within 30 days prior to study drug administration except for the influenza vaccine.
17. Has clinically significant infection (example, pneumonia, pyelonephritis) within 30 days prior to enrollment.
18. Has any unstable or uncontrolled cardiovascular, pulmonary, hepatic, renal, gastrointestinal, genitourinary, hematological, coagulation, immunological, endocrine/metabolic, or other medical disorder that, in the opinion of the investigator, would confound the study results or compromise participant safety.
19. Has had any surgical procedure requiring general anesthesia within 30 days prior to enrollment or is planning to undergo major surgery during the study period.
20. Has any history of malignancy, except for the following: (a) adequately treated nonmetastatic basal cell skin cancer; (b) squamous cell skin cancer that has been adequately treated and that has not recurred for at least 1 year prior to enrollment; and (c) history of cervical carcinoma in situ that has been adequately treated and that has not recurred for at least 3 years prior to enrollment. Participants with remote history of malignancy (example, >10 years since completion of curative therapy without recurrence) will be considered based on the nature of the malignancy and the therapy received and must be discussed with the sponsor on a case-by-case basis prior to enrollment.
21. Has a current or recent history (within 1 year prior to enrollment) of alcohol dependence or illicit drug use.
22. Has active psychiatric problems that, in the investigator's opinion, may interfere with compliance with the study procedures.
23. Is unable to attend all the study visits or comply with study procedures.

    For Part 1 Participants With UC or CD:
24. Has received any investigational or approved biologic or biosimilar agent in the last 6 months prior to Screening.
25. Participant currently requires or is anticipated to require surgical intervention for UC or CD during the study.

    For Part 1 Healthy Participants Only:
26. Has laboratory abnormalities considered to be clinically significant by the investigator during the Screening Period, for example the following:

    * Hemoglobin level less than (<) 10 gram per decilitre (g/dL).
    * White blood cell (WBC) count <3*10^9 per liter (/L).
    * Lymphocyte count <0.5*10^9/L.
    * Platelet count <100*10^9/L or >1200*10^9/L.
    * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >upper limit of normal (ULN).
    * Alkaline phosphatase >ULN.
    * Serum creatinine >1.5*ULN.

    For Part 1 Participants with UC or CD and Part 2 Participants:
27. Has any of the following laboratory abnormalities considered to be clinically significant by the investigator during the Screening Period:

    * Hemoglobin level <8 g/dL.
    * WBC count <3*10^9/L.
    * Lymphocyte count <0.5 x 10^9/L.
    * Platelet count <100*10^9/L or >1200*10^9/L.
    * ALT or AST >3*ULN.
    * Alkaline phosphatase >3*ULN.
    * Serum creatinine >2*ULN.

    For Part 2 only:
28. Has received any investigational or approved biologic or biosimilar agents other than vedolizumab in the last 6 months prior to Screening.
29. The subject has active or latent tuberculosis (TB), this may involve documentation of the participant's TB status prior to commencing vedolizumab with the participant's own treating physician.
30. Has a history of any major neurological disorders, including stroke, multiple sclerosis, brain tumor, or neurodegenerative disease.
31. Has a positive progressive multifocal leukoencephalopathy (PML) subjective symptom checklist at screening and prior to dosing on Day 1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11-01 (Estimated); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
AUCt: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Caffeine | Predose and at multiple time points (up to 24 hours) postdose
AUCt: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Losartan | Predose and at multiple time points (up to 24 hours) postdose
AUCt: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Omeprazole | Predose and at multiple time points (up to 24 hours) postdose
AUCt: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Dextromethorphan | Predose and at multiple time points (up to 24 hours) postdose
AUCt: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Midazolam | Predose and at multiple time points (up to 24 hours) postdose
AUC(0-inf): Area Under the Plasma Concentration-time Curve from Time 0 to Infinity for Caffeine | Predose and at multiple time points (up to 24 hours) postdose
AUC(0-inf): Area Under the Plasma Concentration-time Curve from Time 0 to Infinity for Losartan | Predose and at multiple time points (up to 24 hours) postdose
AUC(0-inf): Area Under the Plasma Concentration-time Curve from Time 0 to Infinity for Omeprazole | Predose and at multiple time points (up to 24 hours) postdose
AUC(0-inf): Area Under the Plasma Concentration-time Curve from Time 0 to Infinity for Dextromethorphan | Predose and at multiple time points (up to 24 hours) postdose
AUC(0-inf): Area Under the Plasma Concentration-time Curve from Time 0 to Infinity for Midazolam | Predose and at multiple time points (up to 24 hours) postdose
Cmax: Maximum Observed Plasma Concentration for Caffeine | Predose and at multiple time points (up to 24 hours) postdose
Cmax: Maximum Observed Plasma Concentration for Losartan | Predose and at multiple time points (up to 24 hours) postdose
Cmax: Maximum Observed Plasma Concentration for Omeprazole | Predose and at multiple time points (up to 24 hours) postdose
Cmax: Maximum Observed Plasma Concentration for Dextromethorphan | Predose and at multiple time points (up to 24 hours) postdose
Cmax: Maximum Observed Plasma Concentration for Midazolam | Predose and at multiple time points (up to 24 hours) postdose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (2):
- United States (2):
  - WCCT, Cypress, California
  - QPS MRA, Miami, Florida